CLINICAL TRIAL: NCT02404922
Title: A Phase I Single Center, Double-Blind, Placebo-Controlled, Multiple Dose-Ascending Study to Evaluate the Pharmacokinetics and Tolerability of CTP-730 Immediate Release at Steady State in Healthy Adults
Brief Title: Multiple Ascending Dose Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CP730.1002
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Safety/Efficacy Study; Randomized; Double Blind

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CTP-730 Low Dose or Matching Placebo (Experimental): Capsule, once daily.
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730
- CTP-730 Mid Dose or Matching Placebo (Experimental): Capsule, once daily
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730
- CTP-730 High Dose or Matching Placebo (Experimental): Capsule, once daily.
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730

INTERVENTIONS:
Drug: CTP-730
Drug: Placebo for CTP-730

SUMMARY:
This study will assess in healthy male and female subjects the safety, tolerability and pharmacokinetics (PK) profiles of Immediate Release CTP-730 at steady state following 7 days of dosing. Three doses of Immediate Release (IR) CTP-730 capsules will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females between 18 and 50 years of age.
* Body weight ≥ 50 kg and BMI within the range of 18 to 30 kg/m2

Exclusion Criteria:

* Medical, psychiatric illness or history of depression that could, in the investigator's opinion, compromise the subject's safety
* Significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
* History of clinically significant central nervous system (eg, seizures), cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal (GI) conditions.
* PR interval ≥ 220 msec or QRS duration ≥ 120 msec or QTcB / QTcF interval > 450 msec obtained at screening visit or prior to the first dose of study drug.
* Liver function tests greater than the upper limit of normal.
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening.
* Urinalysis positive for protein or glucose.
* A positive screen for alcohol, drugs of abuse, or tobacco use.
* Inability to comply with food and beverage restrictions during study participation.
* Donation or blood collection or acute loss of blood prior to screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Profile | 96 hours
  The primary pharmacokinetics parameters of interest will be time to attainment of steady state, and Cmax, Tmax, AUC0-24hr, AUClast and AUCinf at steady state
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 hours
  Adverse events categorized by body system and MedDRA term

CONTACTS AND LOCATIONS:
Overall Officials: Ginny Braman, Study Director — Concert Pharmaceuticals, Inc.
Locations (1):
- CMAX, Adelaide, South Australia, Australia